CLINICAL TRIAL: NCT00728286
Title: Assessment of Platelet-dependent Thrombosis in Patients With Acute Coronary Syndromes Using an ex Vivo Arterial Injury Model
Brief Title: Assessment of Thrombogenicity in Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: British Heart Foundation (Other); University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Other Study IDs: 3639b; British Heart Foundation (Other Grant/Funding Number: FS/033/07)
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus; Acute Coronary Syndrome
Keywords: Type 2 Diabetes Mellitus; Acute Coronary Syndrome; Platelet dependent thrombogenicity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Type 2 diabetes mellitus: We aim to determine the effects of dual antiplatelet therapy with aspirin 75mg once a day and clopidogrel 75mg once a day on platelet dependent thrombogenicity in patients with type 2 diabetes mellitus and acute coronary syndrome. Eighty patients (40 with type 2 diabetes and 40 without) have been studied one week after Non ST-elevation acute coronary syndrome. All patients were on secondary prevention therapy as recommended by international guidelines.

SUMMARY:
The purpose of this study is to assess platelet dependent thrombogenicity in patients after acute coronary syndrome using an ex vivo arterial injury model.

DETAILED DESCRIPTION:
Abnormal platelet activity seen in patients with Type2 Diabetes Mellitus (T2DM) may be an important contributor to their enhanced cardiovascular risk and higher rates of cardiovascular events following acute coronary syndrome, despite dual antiplatelet therapy with aspirin and clopidogrel. We have earlier demonstrated high thrombogenicity in individuals with T2DM and CAD in the absence of acute ischaemic events, despite therapeutic doses of aspirin.We hypothesise that patients with T2DM will have increased thrombogenicity after acute coronary syndrome despite optimal secondary prevention medication.Measuring ex vivo thrombus area using an arterial injury model simulates plaque rupture and reflects the summative effect of all haemostatic abnormalities. The thrombus area of patients with ACS and T2DM will be compared to the controls without T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (WHO criteria) with raised cardiac troponin T
* Aged 18-80 years
* Stable Acute coronary syndrome
* On aspirin and clopidogrel
* Willing to participate in the study

Exclusion Criteria:

* Smoking (current smokers or smokers who quit in the last 6 months preceding recruitment)
* Malignancy (any suspected or proven)
* Haematological disorders (bleeding disorders)
* Pre-menopausal women
* Use of corticosteroids/other antithrombotic agents (warfarin)
* Chronic liver disease
* Unable to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-ST elevation myocardial infarction - Acute Coronary syndrome (ACS) and on existing medication will undergo chamber study
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Thrombus area | Within 10 days after acute coronary syndrome

SECONDARY OUTCOMES:
Factors affecting thrombus area | Within ten days after acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Azfar G Zaman, MD FRCP, Principal Investigator — Freeman Hospital, Newcastle upon Tyne NHS Trust, Newcastle upon Tyne. NE7 7DN
Locations (1):
- Royal Victoria Hospital, Newcastle upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Background] Natarajan A, Marshall SM, Worthley SG, Badimon JJ, Zaman AG. The presence of coronary artery disease increases platelet-dependent thrombosis in patients with type 2 diabetes mellitus. J Thromb Haemost. 2008 Dec;6(12):2210-3. doi: 10.1111/j.1538-7836.2008.03176.x. Epub 2008 Oct 1. No abstract available. PMID 18983525
- [Background] Osende JI, Badimon JJ, Fuster V, Herson P, Rabito P, Vidhun R, Zaman A, Rodriguez OJ, Lev EI, Rauch U, Heflt G, Fallon JT, Crandall JP. Blood thrombogenicity in type 2 diabetes mellitus patients is associated with glycemic control. J Am Coll Cardiol. 2001 Nov 1;38(5):1307-12. doi: 10.1016/s0735-1097(01)01555-8. PMID 11691500
- [Background] Shechter M, Merz CN, Paul-Labrador MJ, Kaul S. Blood glucose and platelet-dependent thrombosis in patients with coronary artery disease. J Am Coll Cardiol. 2000 Feb;35(2):300-7. doi: 10.1016/s0735-1097(99)00545-8. PMID 10676673
- [Background] Helft G, Osende JI, Worthley SG, Zaman AG, Rodriguez OJ, Lev EI, Farkouh ME, Fuster V, Badimon JJ, Chesebro JH. Acute antithrombotic effect of a front-loaded regimen of clopidogrel in patients with atherosclerosis on aspirin. Arterioscler Thromb Vasc Biol. 2000 Oct;20(10):2316-21. doi: 10.1161/01.atv.20.10.2316. PMID 11031221